CLINICAL TRIAL: NCT03409159
Title: Austrian Left Atrial Appendage Closure Registry
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 29-355 ex 16/17
Record Dates: First submitted 2017-11-24; First posted 2018-01-24 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LAAC — Left atrial appendage closure

SUMMARY:
Left atrial appendage (LAA) occlusion (LAAC) has been introduced to treat patients with indication of oral anticoagulation (OAC) for atrial fibrillation (AF) with contraindication to OAC. This registry aims to document all LAAC procedures in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received LAAC in Austria

Exclusion Criteria:

* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation, who received LAAC in Austria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful left atrial appendage closure, as defined by European Society of Cardiology Guidelines | 30 days

SECONDARY OUTCOMES:
Number of participants with death, stroke or bleeding | 5 years
Number of participants with procedure-related adverse events | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No